CLINICAL TRIAL: NCT01349348
Title: A Randomized, Double-blinded, Multicenter, Placebo Controlled, Parallel Designed Study, to Evaluate the Efficacy and Safety of Tolvaptan Tablet in Treatment of Patients With Cirrhosis Ascites, Using Diuretics as Initial Treatment
Brief Title: Phase III Study of Tolvaptan Tablet to Treat Cirrhosis Ascites
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 156-08-805-01
Record Dates: First submitted 2011-05-04; First posted 2011-05-06 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Ascites; Hepatic Cirrhosis
Keywords: Tolvaptan treatment to ascites and hepatic cirrhosis
MeSH Terms: conditions — Ascites; Liver Cirrhosis | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tolvaptan 15mg (Experimental): Tablet;15mg/tab
  Interventions: Drug: Tolvaptan
- Tolvaptan 7.5mg (Experimental): Tablet;7.5mg/tab
  Interventions: Drug: Tolvaptan
- Placebo (Placebo Comparator): Tolvaptan 0mg/tab
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Tolvaptan — tablet, 15 mg, Qd, for 7 days
  Other Names: SAMSCA
  Arms: Tolvaptan 15mg
Drug: Tolvaptan — tablet, 7.5 mg, Qd, for 7 days
  Other Names: SAMSCA
  Arms: Tolvaptan 7.5mg
Drug: placebo — tablet, 7.5/15mg , Qd, 7days.
  Other Names: Blank tablet
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of Tolvaptan 7.5mg and 15mg in treatment of patients with cirrhosis ascites who fail to response adequately to treatment with common diuretics.

DETAILED DESCRIPTION:
For symptoms of fluid retention due to liver diseases (ascites and/or lower extremity edema, i.e. hepatic edema), treatment generally starts with bed rest and a low-salt diet. Aldosterone antagonists and loop diuretics are commonly used diuretics in the treatment of fluid retention due to liver diseases. In aldosterone antagonists' therapy, nevertheless, hyperkalemia is frequently reported, slow onset of action and dose escalation needed also impair its effect. If aldosterone antagonists' therapy is ineffective, loop diuretics as strong diuretics are usually added up. However, Dose escalation of loop diuretics also boost the occurrence of hyponatremia and hypokalemia, and combination of the two drugs provided fastest onset of effectiveness with less adverse events. While, because both diuretics can cause sodium lose which is difficult to prevent and treat, hyponatremia is easy to occur. The combination of aldosterone antagonists and K-sparing diuretics reduces the occurrence of hypokalemia but have little effect on the prevention and treatment of hyponatremia. In addition, there are still some patients who are resistent to loop diuretics or intolerant of an effective diuretic dosage due to adverse events.

Tolvaptan increases the excretion of electrolyte-free water (aquaretic) without changing electrolytes excretion by inhibiting the water reabsorption of collecting duct in kidney. It is demonstrated that Tolvaptan increased urine volume without impairing renal function.

ELIGIBILITY:
Inclusion criteria:

1. Patients diagnosed with liver cirrhosis clinically or pathologically;
2. Patients with ascites confirmed by Type-B ultrasound scan after receiving combination therapies of oral loop diuretics and aldosterone antagonists for at least 4 days with the fixed usage and dosage
3. Inpatients or patients who can be hospitalized for this study from Day -3 (Screening) to Day 8 (the day for efficacy evaluation);
4. Patients with body weight change within ±1.0 kg in the 2 days prior to initiation of treatment (Day -2 and Day -1)
5. Age: 18 to 75 years, inclusive(at the time informed consent is obtained);
6. Genders: men or women;
7. Patients who have signed informed consent form.

Exclusion criteria:

1. Patients with any of the following diseases, complications or symptoms:

   * Hepatic encephalopathy (hepatic coma of grade II or higher1）);
   * Malignant ascites (patients have tumor cells detected in ascites if malignant ascites be highly suspected);
   * Uncontrolled spontaneous bacterial peritonitis;
   * Patients who are likely to experience alimentary tract hemorrhage during the study;
   * Heart failure (NYHA2） grade III or IV);
   * Anuresis (daily urine volume is less than 100mL);
   * Dysuria due to urinary tract stricture, urinary calculus, tumor in the urinary tract or other cause.
2. Patients with history of :

   * Alimentary tract hemorrhage within 10 days prior to screening;
   * Cerebral accident suffered within 30 days prior to screening;
   * Past history of hypersensitivity or idiosyncratic reaction to benzazepine derivatives (Benazepril).
3. Patients with systolic pressure below 90mmHg at screening;
4. Patients with any of the following abnormal laboratory parameters at screening:

   * Serum creatinine >1.5x upper limit of normal range;
   * Serum Na+>145mmol/L (or higher than upper limit of normal range);
   * Serum K+>5.5mmol/L;
5. Patients with Child-pugh score3）>12;
6. Patients who are unable to take medicine orally;
7. Female patients who are pregnant, lactating, or who are at child-bearing age without using acceptable contraceptive means;
8. Patients who received blood products including albumin within 4 days prior to the initiation of treatment
9. Patients who participated in any clinical trial other than tolvaptan within one month prior to screening;
10. Patients who participated in Tolvaptan trials and took Tolvaptan previously;
11. Patients otherwise judged by the investigator, to be inappropriate for inclusion in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2010-10; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in body weight after 7 days randomized treatment (Day 8). | 7 days

SECONDARY OUTCOMES:
Change from baseline in body weight after 4 days randomized treatment (Day 5); | 4days
The rate of change from baseline in body weight after 4, 7 days randomized treatment (Day 5, Day 8); | 4 and 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Minde Zeng, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Tang J, Wang Y, Han T, Mao Q, Cheng J, Ding H, Shang J, Zhang Q, Niu J, Ji F, Chen C, Jia J, Jiang X, Lv N, Gao Y, Wang Z, Wei Z, Chen Y, Zeng M, Mao Y. Tolvaptan therapy of Chinese cirrhotic patients with ascites after insufficient diuretic routine medication responses: a phase III clinical trial. BMC Gastroenterol. 2020 Nov 19;20(1):391. doi: 10.1186/s12876-020-01536-0. PMID 33213378
- [Derived] Wang S, Zhang X, Han T, Xie W, Li Y, Ma H, Liebe R, Weng H, Ding HG. Tolvaptan treatment improves survival of cirrhotic patients with ascites and hyponatremia. BMC Gastroenterol. 2018 Sep 4;18(1):137. doi: 10.1186/s12876-018-0857-0. PMID 30180806